CLINICAL TRIAL: NCT00462345
Title: An Open-label Study to Evaluate the Effect of MabThera in Combination With Methotrexate on Treatment Response in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Anti-TNF Therapies
Brief Title: A Study of MabThera (Rituximab) in Combination With Methotrexate in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to Anti-TNF Therapies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20934
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Adrenal Cortex Hormones; Anti-Inflammatory Agents, Non-Steroidal; Folic Acid

ARMS (1):
- Rituximab, Methotrexate (Experimental): Participants received rituximab 1000 milligrams (mg), intravenously (IV), on Day 1 and Day 15. Participants also received methylprednisolone 100 mg, IV, 30 minutes before the infusion of rituximab. Participants also received methotrexate (MTX) 10 to 25 milligrams per week (mg/week), orally (PO) or parenterally, and folate greater than or equal to (≥) 5 mg/week, PO, folate greater than or equal to (≥) 5 mg/week, PO, either as a single dose or as divided daily doses from Day 1 through Week 24. Participants also received prednisone less than or equal to (≤) 10 milligrams per day (mg/day), PO, OR equivalent corticosteroid, OR non-steroidal anti-inflammatory drugs (NSAIDs), PO, from Day 1 through Week 24. Eligible participants who completed the first 24-week course were entered into a second course.
  Interventions: Drug: rituximab; Drug: Methotrexate; Drug: Corticosteroid or NSAID; Dietary Supplement: Folate

INTERVENTIONS:
Drug: rituximab — 1000 mg i.v. on Days 1 and 15
  Other Names: MabThera; Rituxan
Drug: Methotrexate — 10 to 25 mg/week p.o. or parenteral from Day 1 through Week 24
Drug: Corticosteroid or NSAID — ≤10 mg/day prednisone p.o., or equivalent corticosteroid, or NSAIDs p.o. from Day 1 through Week 24
Dietary Supplement: Folate — ≥5 mg/week, once daily or b.i.d. from Day 1 through Week 24

SUMMARY:
This single arm study will evaluate the efficacy and safety of MabThera in combination with methotrexate in patients with rheumatoid arthritis who have had an inadequate response to one or more anti-TNF therapies. Patients will receive MabThera 1000mg i.v. on days 1 and 15, and methotrexate (10-25mg/week p.o. or parenteral), together with methylprednisolone 100mg i.v. prior to infusion of MabThera. After week 24, eligible patients may receive re-treatment. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-80 years of age;
* rheumatoid arthritis for >=6 months;
* receiving outpatient treatment;
* an inadequate response to at least one anti-TNF therapy;
* stable methotrexate for >=12 weeks.

Exclusion Criteria:

* other rheumatic autoimmune disease or inflammatory joint disease;
* previous treatment with MabThera;
* concurrent treatment with any DMARD (apart from methotrexate), anti-TNF alpha therapy, or other biologic agent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Vieira MC, Zwillich SH, Jansen JP, Smiechowski B, Spurden D, Wallenstein GV. Tofacitinib Versus Biologic Treatments in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Tumor Necrosis Factor Inhibitors: Results From a Network Meta-analysis. Clin Ther. 2016 Dec;38(12):2628-2641.e5. doi: 10.1016/j.clinthera.2016.11.004. Epub 2016 Nov 24. PMID 27889300

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab, Methotrexate: Participants received rituximab 1000 milligrams (mg), intravenously (IV), on Day 1 and Day 15; methylprednisolone 100 mg, IV, was administered 30 minutes before each infusion of rituximab. Participants also received methotrexate (MTX) 10 to 25 milligrams per week (mg/week), orally (PO) or parenterally, and folate at a stable dose of greater than or equal to (≥) 5 mg/week, PO, either as a single dose or as divided daily doses from Day 1 through Week 24. Participants also received prednisone less than or equal to (≤) 10 milligrams per day (mg/day), PO, OR equivalent corticosteroid, OR non-steroidal anti-inflammatory drugs (NSAIDs), PO, from Day 1 through Week 24. Eligible participants who completed the first 24-week course were entered into a second course.
Period: Overall Study
Arm/Group | Rituximab, Methotrexate
Started | 40
Completed First Course | 38
Completed | 37
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Did not complete second course | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all enrolled participants who received the investigational treatment.
Groups:
- Rituximab, Methotrexate: Participants received rituximab 1000 mg, IV, on Day 1 and Day 15; methylprednisolone 100 mg, IV, was administered 30 minutes before each infusion of rituximab. Participants also received MTX 10 to 25 mg/week, PO or parenterally, and folate at a stable dose of ≥5 mg/week, PO, either as a single dose or as divided daily doses from Day 1 through Week 24. Participants also received prednisone ≤10 mg/day, PO, OR equivalent corticosteroid, OR NSAIDs, PO, from Day 1 through Week 24. Eligible participants who completed the first 24-week course were entered into a second course.
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With An American College of Rheumatology 20 Percent (%) Improvement Criteria (ACR20) Response at Week 24
Description: ACR20 response: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 of 5 remaining ACR core measures: Patient Assessment of Pain; Patient Global Assessment of Disease Activity (PtGA); Physician Global Assessment of Disease Activity (PGA); self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ-DI]); and either C-Reactive Protein (CRP) or erythrocyte sedimentation rate (ESR).
Time Frame: Week 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
percentage of participants | 47.5 [31.5 to 63.9]

2. Secondary Outcome: Percentage of Participants With An American College of Rheumatology 50% Improvement Criteria (ACR50) Response at Week 24
Description: ACR50 response: ≥50% improvement in tender joint count; ≥50% improvement in swollen joint count; and ≥50% improvement in at least 3 of 5 remaining ACR core measures: Patient Assessment of Pain; PtGA; PGA; self-assessed disability (HAQ-DI); and either CRP or ESR.
Time Frame: Week 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
percentage of participants | 7.5 [1.6 to 20.4]

3. Secondary Outcome: Percentage of Participants With An American College of Rheumatology 70% Improvement Criteria (ACR70) Response at Week 24
Description: ACR70 response: ≥70% improvement in tender joint count; ≥70% improvement in swollen joint count; and ≥70% improvement in at least 3 of 5 remaining ACR core measures: Patient Assessment of Pain; PtGA; PGA; self-assessed disability (HAQ-DI); and either CRP or ESR.
Time Frame: Week 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
percentage of participants | 5.0 [0.6 to 16.9]

4. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS-28)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (millimeters per hour [mm/hr]) and PtGA of disease activity with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 ≤3.2 equals (=) low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
scores on a scale
  Week 0 | 6.76 (1.02)
  Week 24 | 5.31 (1.16)
  Change at Week 24 | -1.45 (0.94)

5. Secondary Outcome: Percentage of Participants With Change in DAS-28 From BL to Week 24 of ≥1.2
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (mm/hr) and PtGA of disease activity with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity.
Time Frame: Baseline, Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
percentage of participants | 60.0

6. Secondary Outcome: Percentage of Participants With DAS Response by European League Against Rheumatism (EULAR) Category at Week 24
Description: The percentage of participants categorized as good, moderate, or nonresponders according to the EULAR response criteria at Week 24. Participants were categorized as good responders if the intensity of their symptoms was in the "low disease activity (DAS28 less than [<]3.2)" category after treatment, and their symptoms significantly decreased to >1.2. Participants were categorized as moderate responders if the intensity of their symptoms was in the "moderate or high disease activity (DAS28 >3.2)" category after treatment, and the symptoms significantly decreased to >1.2; or if the intensity of their symptoms was in the "low or moderate disease activity (DAS28 <5.1)" category, and the DAS28 score changed more than 0.6 or 1.2 or less. Participants were categorized as non-responders if they did not fall into the good or moderate categories.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
percentage of participants
  Good responders | 5.0
  Moderate responders | 65.0
  Nonresponders | 30.0

7. Secondary Outcome: Swollen Join Count (SJC)
Description: Number of swollen joints was determined by examination of 66 joints (as assessed through pressing and palpating during the physical examination) and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit as swollen or not swollen.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
swollen joints
  Week 0 | 16.3 (8.4)
  Change at Week 24 | -8.9 (6.2)
  Change at Week 48 | -11.6 (7.2)

8. Secondary Outcome: Tender Joint Count (TJC)
Description: Number of tender joints was determined by examination of 68 joints (as assessed through pressing and palpating during the physical examination) and identifying when swelling was present. The number of tender joints was recorded on the joint assessment form at each visit as either tender or not tender.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
tender joints
  Week 0 | 21.9 (14.0)
  Change at Week 24 | -9.0 (9.3)
  Change at Week 48 | -13.9 (11.1)

9. Secondary Outcome: Patient Global Assessment of Disease Activity (VAS)
Description: The mean score of the symptoms of rheumatoid arthritis (RA) at Week 0 (baseline) and the change from Week 0 to Weeks 24 and 48 as assessed by participants using a 100 mm horizontal VAS, where the left endpoint indicated "No disease activity" (no symptom, or no symptom of RA), and the right endpoint indicated "Maximum disease activity" (maximum RA activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
mm
  Week 0 | 72.6 (21.6)
  Change at Week 24 | -20.5 (25.8)
  Change at Week 48 | -31.8 (26.9)

10. Secondary Outcome: Physician Global Assessment of Disease Activity (VAS)
Description: The mean score of the symptoms of RA at Week 0 and the change from Week 0 (baseline) to Weeks 24 and 48 as assessed by investigators using a 100-mm horizontal VAS, where the left endpoint indicated "No disease activity" (no symptom, or no symptom of RA), and the right endpoint indicated "Maximum disease activity" (maximum RA activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
mm
  Week 0 | 72.8 (13.4)
  Change at Week 24 | -30.4 (24.1)
  Change at Week 48 | -42.1 (23.0)

11. Secondary Outcome: Patient Assessment of Pain (VAS)
Description: The mean score of pain at Week 0 (baseline) and the change from Week 0 to Weeks 24 and 48 as assessed by participants using a 100-mm horizontal VAS, where the left endpoint indicated "No pain," and the right endpoint indicated "Unbearable pain." A negative change indicated improvement.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
mm
  Week 0 | 69.3 (20.7)
  Change at Week 24 | -16.8 (26.1)
  Change at Week 48 | -28.2 (26.8)

12. Secondary Outcome: C-reactive Protein (CRP) Level
Description: The mean level of CRP in milligrams per liter (mg/L), an acute phase reactant, at Week 0 and the change from Week 0 to Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
mg/L
  Week 0 | 3.80 (4.32)
  Change at Week 24 | -1.54 (3.85)
  Change at Week 48 | -2.23 (3.01)

13. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: The mean level of ESR (in mm/hr), an acute phase reactant, at Week 0 and the change from Week 0 to Weeks 24 and 48.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
mm/hr
  Week 0 | 77.2 (28.6)
  Change at Week 24 | -23.4 (27.1)
  Change at Week 48 | -36.1 (26.0)

14. Secondary Outcome: HAQ-DI Score
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 40
scores on a scale
  Week 0 | 1.66 (0.70)
  Change at Week 24 | -0.34 (0.58)
  Change at Week 48 | -0.53 (0.64)

15. Secondary Outcome: Physical Function as Assessed by Short Form 36 (SF-36)
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Screening, Weeks 24 and 48
Population: ITT population; n (number) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 39
scores on a scale
  Screening, Physical functioning (n=39) | 27.7 (17.2)
  Screening, Role-physical (n=39) | 26.6 (21.5)
  Screening, Bodily pain (n=39) | 29.2 (17.5)
  Screening, General health (n=39) | 31.7 (16.2)
  Week 24, Physical functioning (n=39) | 35.8 (22.5)
  Week 24, Role-physical (n=39) | 41.5 (23.1)
  Week 24, Bodily pain (n=39) | 44.7 (19.7)
  Week 24, General health (n=39) | 38.1 (17.1)
  Week 48, Physical functioning (n=39) | 43.4 (26.7)
  Week 48, Role-physical (n=38) | 49.3 (29.0)
  Week 48, Bodily pain (n=38) | 50.9 (22.7)
  Week 48, General health (n=38) | 44.9 (22.7)

16. Secondary Outcome: SF-36 Mental Component Scores
Description: as for outcome 15
Time Frame: Screening, Weeks 24 and 48
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 39
scores on a scale
  Screening, Vitality (n=38) | 30.3 (18.6)
  Screening, Social functioning (n=39) | 41.7 (26.8)
  Screening, Role-emotional (n=39) | 36.8 (25.3)
  Screening, Mental health (n=38) | 52.9 (19.5)
  Week 24, Vitality (n=39) | 35.7 (21.2)
  Week 24, Social functioning (n=39) | 55.5 (25.6)
  Week 24, Role-emotional (n=39) | 53.9 (27.6)
  Week 24, Mental health (n=39) | 56.0 (21.4)
  Week 48, Vitality (n=38) | 44.2 (26.6)
  Week 48, Social functioning (n=38) | 63.2 (26.0)
  Week 48, Role-emotional (n=38) | 55.5 (31.9)
  Week 48, Mental health (n=38) | 60.7 (23.9)

17. Secondary Outcome: Modified Total Sharp-Genant Score (mTSS)
Description: Posterior-anterior (PA) radiograph of each hand and anterior-posterior (AP) radiograph of each foot were taken separately and assessed according to Genant's method as modified from Sharp's method. The Sharp-Genant score=total of the erosion score and the joint space narrowing (JSN) score of all the hands and feet. Erosion Score: 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. JSN Score:13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). Maximum total erosion score in hands=100 and in feet=42; maximum scores for JSN in the hands=100 and in feet=48. Maximum modified Sharp score achievable is 290. A lower number change from Baseline indicated a better score. Change in scores was calculated as change=final score minus initial score.
Time Frame: Screening and Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 39
scores on a scale
  Screening | 79.5 (48.5)
  Change at Week 24 | 0.26 (0.55)
  Change at Week 48 | 0.64 (1.16)

18. Secondary Outcome: Modified Sharp Radiographic Erosion Score (ES)
Description: Erosion Score: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. Maximum total erosion score in the hands was 100 and in the feet was 42, for a maximum overall score of 142. Total erosion score was for both hands and feet.
Time Frame: Screening, Weeks 24 and 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 39
scores on a scale
  Screening | 25.2 (25.1)
  Change at Week 24 | 0.18 (0.42)
  Change at Week 48 | 0.49 (0.89)

19. Secondary Outcome: Modified Sharp Radiographic Joint Space Narrowing Score (JSN)
Description: JSN Score: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). Maximum total scores for JSN in the hands was 100 and in the feet was 48, for a maximum overall score of 148. Total JSN was for both hands and feet.
Time Frame: Screening, Weeks 24 and 48
Population: ITT population. 39 participants were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab, Methotrexate
Number analyzed (Participants) | 39
scores on a scale
  Screening | 54.3 (27.6)
  Change at Week 24 | 0.08 (0.24)
  Change at Week 48 | 0.15 (0.51)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from Screening up through Week 48 or Withdrawal Visit.
Description: All enrolled participants who received study treatment were included in the safety analysis. The study did not include a separate analysis of nonserious AEs, therefore AEs presented in this record include all AEs reported during the study, not just nonserious events.
Arm/Group | Rituximab, Methotrexate
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab, Methotrexate (N=40)
Appendicitis (Gastrointestinal disorders) | 2
Arthritis bacterial (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Scrub typhus (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab, Methotrexate (N=40)
Upper respiratory tract infection (Infections and infestations) | 12
Onychomycosis (Infections and infestations) | 3
Appendicitis (Infections and infestations) | 2
Arthritis bacterial (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Scrub typhus (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Urticaria (Musculoskeletal and connective tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Feeling hot (General disorders) | 4
Chest discomfort (General disorders) | 2
Face oedema (General disorders) | 2
Pyrexia (General disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Irritability (General disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Amnesia (Nervous system disorders) | 2
Disturbance in attention (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Neck injury (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Breast mass (Reproductive system and breast disorders) | 1
Galactorrhoea (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Iridocyclitis (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Blood pressure decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Vasculitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.